CLINICAL TRIAL: NCT03666624
Title: Socially Isolated Older Adults Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Hyun-Jun Kim, Research Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005149; 5P30AG034592-05 (NIH)
Record Dates: First submitted 2018-09-07; First posted 2018-09-12 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Alzheimer Disease; Dementia
Keywords: LGBT
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: This study will utilize a 2-group randomized controlled trial design including 2 assessments, i.e. a pre-treatment and a post-treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized care network (Experimental): 9 60-minute virtual sessions for 6 weeks plus personalized exercise coaching once a week for 6 weeks
  Interventions: Behavioral: Personalized care network
- Routine medical care (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Personalized care network — The Personalized care network intervention includes exercise training for participant with dementia and behavioral management training for addressing challenges.
  Arms: Personalized care network

SUMMARY:
The lack of efficacious research-based interventions for sexual and gender minority (SGM) older adults living with Alzheimer's disease and other dementias, combined with the heightened risk of cognitive impairment in this population, presents a significant public health problem. SGM older adults are at elevated risk of social isolation and experience significant barriers to healthcare access. Existing interventions for older adults with dementia have been found to be effective for caregiving dyads. Yet SGM older adults, compared to heterosexuals, are significantly less likely to be married or to have biological family members to support them. A significant proportion of SGM older adults living with dementia have no caregiver or care network. The goal of the proposed research is to design and pilot test the cultural appropriateness, acceptability, and feasibility of an innovative translation of a personalized care network-RDAD (Reducing Disability in Alzheimer's Disease) to support those living with dementia without a family caregiver, directly addressing unique SGM-specific risk factors.

DETAILED DESCRIPTION:
We will address the following aims:

Aim 1. Develop a personalized care network-RDAD intervention suitable for SGM older adults living with dementia without caregivers.

Aim 2. Implement a preliminary randomized controlled trial (RCT) of 30 participants with 2 arms (routine medical care vs. the personalized care network-RDAD approach) to assess the acceptability, feasibility, and initial efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment is 50 years of age or older
* Self-identify as LGBT (or sexual or gender non-binary or same sex sexual behavior)
* Have early stage dementia, including Alzheimer's disease or needs help with complex daily activities
* Living in the community, not in a care facility.

Exclusion Criteria:

* Known terminal illness (with death anticipated within the next 12 months)
* Hospitalization for a psychiatric disorder in the 12 months prior to baseline
* Have more than early stage dementia
* Any physical limitations/chronic conditions preventing participation in an exercise program.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Jun Kim, PhD, Study Director — University of Washington
Locations (1):
- UWashington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Personalized Care Network | Routine Medical Care
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — participant grieving over recent death of parent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Care Network | Routine Medical Care | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (1.8) | 68.8 (2.0) | 68.6 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 11 | 21
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity
Description: Minutes spent on exercising per week in the past month were calculated from the following two questions: (1) How much time did you spend on exercises (hours per day) on a typical day during the last month; (2) How many days did you spend on exercises during the last month.
Time Frame: Baseline (pre-treatment) and 7 weeks (post-treatment)
Measure: Mean (Standard Error); unit: minutes per week
Arm/Group | Personalized Care Network | Routine Medical Care
Number analyzed (Participants) | 14 | 15
minutes per week
  Unadjusted mean at baseline | 227 (69) | 282 (129)
  Unadjusted mean at 7 weeks | 380 (105) | 232 (76)

2. Primary Outcome: Change in Physical Functioning
Description: Physical Functioning subscale of the Medical Outcomes Study 36-Item Short Form (SF-36) consists of 10 items and measures how much participants' health status limits their activities including walking, climbing, lifting, and bathing or dressing oneself, based on self-reports. Each item is measured a 3-point scale (1 = Yes, limited a lot; 2 = Yes, limited a little; 3 = No, not limited at all), then recoded into 0, 50, and 100, respectively. The recoded scores are averaged to generate a summary score with its possible range from 0 to 100. Higher scores indicate better physical functioning.
Time Frame: Baseline (pre-treatment) and 7 weeks (post-treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Personalized Care Network | Routine Medical Care
Number analyzed (Participants) | 14 | 15
score on a scale
  Unadjusted score at baseline | 66.1 (6.7) | 73.0 (6.1)
  Unadjusted score at 7 weeks | 73.2 (7.3) | 72.0 (6.2)

3. Secondary Outcome: Change in Quality of Life
Description: Quality of Life in Alzheimer's Disease (QOL-AD) is a 13-item scale that measures participant's self-reported feelings about different aspects of life including energy, mood, living situation, memory, family, friends, ability, and money. Each item has a 4-point response scale (1 = poor; 2 = fair; 3 = good; 4 = excellent). The summary score is a sum of the 13 items with its possible range from 13 to 52. Higher scores indicate higher quality of life.
Time Frame: Baseline (pre-treatment) and 7 weeks (post-treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Personalized Care Network | Routine Medical Care
Number analyzed (Participants) | 14 | 15
score on a scale
  Unadjusted score at baseline | 30.9 (2.3) | 32.2 (1.8)
  Unadjusted score at 7 weeks | 32.7 (3.3) | 32.0 (1.5)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Personalized Care Network | Routine Medical Care
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT03666624/Prot_SAP_000.pdf